CLINICAL TRIAL: NCT06232850
Title: Examining the Relationship Between Wrist Position Sense and Manual Dexterity in Individuals With Multiple Sclerosis
Brief Title: Wrist Position Sense in Individuals With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, müge içelli, lecturer, Pamukkale University
Other Study IDs: PU-FTR-MI-02
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Manual Dexterity; Position Sense
MeSH Terms: conditions — Multiple Sclerosis | interventions — Proprioception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple sclerosis patient: According to EDSS should be between 0-3, not having had an attack in the last 3 months and without spasticity according to MAS in patient with MS will assesment KFORCE Sens® device and Purdue Pegboard Test.
  Interventions: Other: Position sense and manual dexterity evaluate
- Healthy group: Healthy people of similar age who agree to participate in the study will evaluate the KFORCE Sens® device and the Purdue Pegboard Test.
  Interventions: Other: Position sense and manual dexterity evaluate

INTERVENTIONS:
Other: Position sense and manual dexterity evaluate — Position sense and manual dexterity evaluate

SUMMARY:
No study has been found examining the effect of wrist position sense on manual dexterity in individuals with multiple sclerosis.The purpose of this study is to examine the effect of wrist position sense on manual dexterity of the hand.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic demyelinating disease of the central nervous system that occurs in young adults and usually progresses with attacks and remissions. As the disease progresses, symptoms such as fatigue, muscle weakness, loss of balance, loss of sensation, spasticity, visual disturbances and bladder dysfunction are observed. In addition to these symptoms, hand functions may be affected even in the early stages of the disease.

Appropriate motor control and mobility skills are required to perform manual dexterity effectively. Joint stabilization and perception of the joint's position and movement in space are needed for motor control of hand functions. In this process, position sense signals contribute significantly to the target localization and performance of the hand. Position sense signals must be constantly updated for the coordination and integration of hand position during manual activities such as holding or grasping an object. This is possible with a healthy sense of position.

Although it is known that position sense is affected in MS patients, no study has been found examining the effect of wrist position sense on manual dexterity. The purpose of this study is to examine the effect of wrist position sense on hand dexterity. Patients' manual dexterity will be evaluated using the Purdue Pegboard Test, and wrist position sense will be evaluated using the K-FORCE Sens® electrogoniometer.

ELIGIBILITY:
Inclusion Criteria:

* Patient group:

  * Disability score (EDSS: Expanded Disability Status Scale) should be between 0-3.
  * Being between the ages of 18-50
  * Not having had an attack in the last 3 months
  * Scoring 24 points or above on the Mini-Mental State Examination
  * Patients diagnosed with relapsing-remitting MS with a disease duration of at least 2 years
  * Patients without spasticity according to MAS

Control group:

* Volunteers in a similar age range who agreed to participate in the study
* Being between the ages of 18-50

Exclusion Criteria:

* Patient group:

  * Presence of diagnosed visual impairment
  * Having other chronic diseases not related to MS
  * Having any orthopedic, neurological, rheumatological or metabolic diagnosis that causes upper extremity involvement
  * History of hand and upper extremity disorders, peripheral nerve disorders, and medical or psychiatric disorders that may significantly affect cognitive function
  * Presence of wrist joint range of motion limitation

Control group:

* Having any orthopedic, neurological, rheumatological or metabolic diagnosis that causes upper extremity involvement
* History of hand and upper extremity disorders, peripheral nerve disorders, and medical or psychiatric disorders that may significantly affect cognitive function
* Presence of wrist joint range of motion limitation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: MS and healthy individuals who proper the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Wrist Position Sense Assessment | four mounth
  Wrist position sense will be assessed with the KFORCE Sens® electrogoniometer. Target measurement values of 30° for wrist flexion, 30° for extension, 10° for radial deviation and 15° for ulnar deviation will be used.

SECONDARY OUTCOMES:
Purdue Pegboard Test (PPT) | four mounth
  PPT evaluates the gross motor skills of the arm, hand and fingers, as well as the fine motor skills of the fingers and fingertips, both unilaterally and bilaterally. It consists of pins, washers, nuts and assembly tests. The test consists of 5 sub-steps (inserting pins with the dominant/non-dominant hand/both hands, mathematical summation and assembly). The scoring of the test is the total number of pins, washers and nuts installed at the end of the given period. One trial will be made for each subtest.

CONTACTS AND LOCATIONS:
Overall Officials: Müge İçelli Güneş, M.Sc., Principal Investigator — Pamukkale University Denizli Health Services Vocational School of Higher Education
Locations (1):
- Müge içelli güneş, Denizli, Deni̇zli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No